CLINICAL TRIAL: NCT01593410
Title: A Multi-center, Open-Label Phase II Study to Determine the Efficacy and Safety of Lenalidomide Plus Low-Dose Dexamethasone in Chinese Subjects With Relapsed/Refractory Multiple Myeloma
Brief Title: Study of Lenalidomide and Low-Dose Dexamethasone in Chinese Subjects With Relapsed/Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-MM-021
Record Dates: First submitted 2012-05-04; First posted 2012-05-08 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Multiple Myeloma
Keywords: Efficacy/Safety; Lenalidomide and Low-Dose Dexamethasone; Chinese Subjects; Relapsed/Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lenalidomide and dexamethasone (Experimental): Cycle 1: 25 mg oral lenalidomide once daily on Days 1-21 every 28 Days and 40 mg oral dexamethasone on Days 8, 15, and 22. Cycle 2 and beyond: 25 oral lenalidomide once daily on Days 1-21 every 28 days and 40 mg oral dexamethasone once daily on Days 1, 8, 15, and 22.
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Lenalidomide — 25 mg oral lenalidomide once daily on Days 1-21 every 28 days
  Other Names: Revlimid
Drug: Dexamethasone — Cycle 1: 40 mg oral dexamethasone once daily on Days 8, 15, and 22. Cycle 2 and beyond: 40 mg oral dexamethasone once daily on Days 1, 8, 15, and 22

SUMMARY:
The purpose of this study is to determine the efficacy of lenalidomide plus low-dose dexamethasone in Chinese subjects with relapsed or refractory multiple myeloma.

Even though the efficacy and safety of lenalidomide has already been well-demonstrated in other populations including Asians, this study will assess the efficacy and safety as well as pharmacokinetics of lenalidomide in Chinese subjects. In addition, this study will generate clinically meaningful information in guiding the therapeutic use of lenalidomide for Chinese subjects.

DETAILED DESCRIPTION:
This is a Phase II, multicenter, single arm, open-label trial which will enroll Chinese subjects in China with relapsed/refractory multiple myeloma that will assess the efficacy and safety of lenalidomide plus low-dose dexamethasone regimen (Rd) given until progressive disease (PD) or discontinuation of lenalidomide for any reason.

There are two cohorts in this protocol, Pharmacokinetic Assessment Treatment Cohort and Treatment Cohort without Pharmacokinetic (PK) Assessment. The first 10 subjects who are ≤ 75 years old and have a baseline Creatinine Clearance ≥ 60 mL/min will participate in pharmacokinetic assessment during the first 8 days of Cycle 1. During this cohort, all subjects will receive 25mg oral lenalidomide once daily on days 1 -21 of each 28-day cycle. During the first cycle of this cohort, subjects will also receive 40mg oral dexamethasone daily on Days 8, 15, and 22 (and no dexamethasone on day 1). Beginning with Cycle 2, subjects will receive 25mg oral lenalidomide once daily on days 1 -21 of each 28-day cycle and 40mg oral dexamethasone daily on Days 1, 8, 15 and 22 of each 28-day cycle.

Once 10 subjects have been enrolled in the PK Assessment Treatment Cohort, the Treatment Cohort without PK Assessment will begin. During this cohort, subjects will receive lenalidomide 25 mg p.o. once daily on Days 1-21 and dexamethasone 40 mg p.o. once daily on Days 1, 8, 15, and 22 of each 28-day cycle. In both cohorts, subjects will continue Rd therapy until the documentation of PD or discontinuation of study therapy due to any reason including intolerable toxicity.

For the primary analysis, response will be assessed according to the European Group for Blood and Marrow Transplantation EBMT (Bladé) criteria by an Independent Response Adjudication Committee (IRAC). Response will also be assessed according to the International Myeloma Working Group (IMWG) criteria and used as an exploratory analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign informed consent form
2. Age ≥ 18 years at the time of signing consent
3. Prior or current diagnosis of Durie-Salmon Stage II or III multiple myeloma AND have disease progression after at least 2 cycles of systemic anti-myeloma treatment or have relapsed with progressive disease after treatment.
4. Measurable levels of myeloma paraprotein in serum (≥ 0.5 g/dL [5 g/L] or urine (≥ 0.2 g excreted in a 24-hour collection sample).
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
6. Able to adhere to the study visit schedule and other protocol requirements.
7. Must agree to comply to Lenalidomide Pregnancy Prevention Risk Management Plan requirements.

Exclusion Criteria

1. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
2. Subjects with non-secretory multiple myeloma by Serum Protein Electrophoresis (SPEP) and Urine Protein Electrophoresis (UPEP) assessment.
3. Pregnant or lactating females
4. Any of the following laboratory abnormalities:

   * Absolute neutrophil count of < 1000 cells/mm3 (1.0 X 109/L)
   * Platelet count < 50,000/mm3 (50 X 109/L) in subjects in whom < 50% of the bone marrow nucleated cells were plasma cells
   * Renal failure requiring dialysis or peritoneal dialysis
   * Serum glutamic oxaloacetic transaminase, (SGOT)/ Aspartate-Aminotransferase (AST) > 3.0 x upper limit of normal (ULN)
   * Serum total bilirubin > 2.0 mg/dL (34μmol/L)
5. Any condition, including the presence of laboratory abnormalities, which placed subject at unacceptable risk if participating in the study or which would confound the ability to interpret study data.
6. Significant active cardiac disease within the previous 6 months.
7. Prior history of malignancies, other than multiple myeloma, unless the subject has been free of disease for ≥ 3 years. Exceptions include the following:

   * Basal cell carcinoma of the skin
   * Carcinoma in situ of the cervix
   * Carcinoma in situ of the breast
   * Squamous cell carcinoma of the skin
8. Incidental histologic finding of prostate cancer (Tumor, Node, and Metastasis [TNM] stage of T1a or T1b)
9. Known hypersensitivity to thalidomide or dexamethasone
10. Prior history of uncontrollable side effects to dexamethasone therapy
11. Peripheral neuropathy ≥ grade 2
12. Prior use of lenalidomide
13. Use of any standard/experimental anti-myeloma drug therapy within 28 days of the start of study drug or use of any experimental non-drug therapy (e.g. donor leukocyte/mononuclear cell infusion) within 56 days of the start of study drug)
14. Unable or unwilling to undergo antithrombotic therapy
15. History of deep vein thrombosis (DVT) or pulmonary emboli (PE) within the past 12 months
16. Known HIV positivity
17. Active infectious hepatitis A, B, or C or chronic carriers of hepatitis B with hepatitis B surface antigen (HBsAG) positive or if the hepatitis B viral deoxyribonucleic acid (HBV DNA) level is detectable by polymerase chain reaction (PCR).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2010-08-01 (Actual); Primary Completion 2013-01-03 (Actual); Study Completion 2013-01-03 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | Up to 24 months
  Complete Response (CR) or partial Response (PR) using the European Group for Blood and Marrow Transplantation (EBMT) (Bladé) criteria.

SECONDARY OUTCOMES:
Adverse Events | Up to 24 months
  Number of participants with Adverse Events
Progression Free Survival (PFS) | Up to 24 months
  Number of participants who survive without progressing by the EBMT (Bladé) criteria
Overall Survival | Up to 24 months
  Number of participants alive
Response duration | Up to 24 months
  Length of time participants respond
Maximum observed concentration in plasma | Days 1, 2, 7, 8, and 9 of Cycle 1
  Pharmacokinetics - Cmax
Area under the plasma concentration-time curve | Days 1, 2, 7, 8, and 9 of Cycle 1
  Pharmacokinetics - AUC
Time to maximum concentration | Days 1, 2, 7, 8, and 9 of Cycle 1
  PK- Tmax
Terminal half-life | Days 1, 2, 7, 8, and 9 of Cycle 1
  Pharmacokinetics - T1/2
Apparent total body clearance | Days 1, 2, 7, 8, and 9 of Cycle 1
  Pharmacokinetics - CL/F
Apparent volume of distribution | Days 1, 2, 7, 8, and 9 of Cycle 1
  Pharmacokinetics - Vz/F

CONTACTS AND LOCATIONS:
Overall Officials: Jay Mei, M.D., Study Director — Celgene
Locations (12):
- China (12):
  - 307 Hospital of Chinese PLA, Beijing
  - Peking University Third Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Chinese PLA General Hospital, Beijing
  - Xiangya Hospital of Central- South University, Changsha
  - Guangdong General Hospital, Guangzhou
  - Nanfang Hospital of Southern Medical University, Guangzhou
  - The First Hospital Affiliated of College Medicine, Zhejiang University, Hangzhou
  - Shanghai Changzheng Hospital, Shanghai
  - Shanghai 6th People's Hospital, Shanghai
  - Changhai Hospital, Shanghai
  - The First Affiliated Hospital of Soochow University, Suzhou

REFERENCES:
- [Background] Hou J, Du X, Jin J, Cai Z, Chen F, Zhou DB, Yu L, Ke X, Li X, Wu D, Meng F, Ai H, Zhang J, Wortman-Vayn H, Chen N, Mei J, Wang J. A multicenter, open-label, phase 2 study of lenalidomide plus low-dose dexamethasone in Chinese patients with relapsed/refractory multiple myeloma: the MM-021 trial. J Hematol Oncol. 2013 Jun 19;6:41. doi: 10.1186/1756-8722-6-41. PMID 23782711
- See also: Link to CSR synopsis — http://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/clinical-study-report-csr-synopses/purposes-of-posting-clinical-study-report-csr-synopses